CLINICAL TRIAL: NCT03147859
Title: Vedolizumab Treatment in Antiretroviral Drug Treated Chronic HIV Infection
Acronym: HAVARTI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Cheo Research Institute (Other); Nebraska Centre for Substance Abuse Research (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20160928-01H
Record Dates: First submitted 2017-04-03; First posted 2017-05-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: HIV-infection/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A-150mg dose of vedolizumab per infusion followed by ATI - Low Dose (Experimental): * Please note that the previous low dose arm was 75mg of vedolizumab per infusion, but no participant was ever given this dose. The study will have a 20-week treatment phase and a 28-week follow-up phase over one year. Intravenous infusion of 150 mg of vedolizumab per infusion per visit schedule will be administered to 4 participants. The visit schedule will be the same for each group - Infusion at weeks 0, 2, 5, 8 and every 4 weeks thereafter up to 40 weeks for at least 7 doses as tolerated. ATI will begin between weeks 6 and 7, and infusions continued at weeks 8, 12, 16 and 20.
  Interventions: Biological: Vedolizumab (brand name Entyvio)
- Group B-300mg dose of vedolizumab per infusion followed by ATI - Mid Dose (Experimental): The study will have a 20-week treatment phase and a 28-week follow-up phase over one year. Intravenous infusion of 300 mg of vedolizumab per infusion per visit schedule will be administered to 4 participants. The visit schedule will be the same for each group - Infusion at weeks 0, 2, 5, 8 and every 4 weeks thereafter up to 40 weeks for at least 7 (and up to 12) doses as tolerated. ATI will begin between week 10, and infusions continued at weeks 12, 16 and 20. Infusions may also be given at weeks 24, 28, 32, 36 and 40 depending on tolerance and pVL response.
  Interventions: Biological: Vedolizumab (brand name Entyvio)
- Group C-600mg dose of vedolizumab per infusion followed by ATI - High Dose (Experimental): The study will have a 20-week treatment phase and a 28-week follow-up phase over one year. Intravenous infusion of 600 mg of vedolizumab per infusion per visit schedule will be administered to 4 participants. The visit schedule will be the same for each group - Infusion at weeks 0, 2, 5, 8 and every 4 weeks thereafter up to 40 weeks for at least 7 (and up to 12) doses as tolerated. ATI will begin between week 10, and infusions continued at weeks 12, 16 and 20. Infusions may also be given at weeks 24, 28, 32, 36 and 40 depending on tolerance and pVL response.
  Interventions: Biological: Vedolizumab (brand name Entyvio)

INTERVENTIONS:
Biological: Vedolizumab (brand name Entyvio) — IV infusion

SUMMARY:
Background:

In nearly all people with human immunodeficiency virus (HIV) infection, immunity cannot either control or eradicate the infection. There are good medicinal treatments, collectively called "ART" (antiretroviral therapy) which control HIV infection by suppressing the virus in the bloodstream. ART is needed for life, and if a person stops taking ART the HIV infection returns in the bloodstream. So, there is good treatment, but no cure. The researchers want to test whether a period of treatment with vedolizumab can be used to control HIV infection in the bloodstream in persons with HIV on ART, after stopping ART.

Objective:

To determine whether vedolizumab is safe and tolerable in people with HIV, to assess the safety of an analytical treatment interruption (ATI), and to determine whether vedolizumab can control HIV infection in the bloodstream without the use of ART.

Eligibility:

Adults 18-65 with HIV who are being treated with ART

Design:

Participants will be screened with: Physical exam, medical history, blood and urine tests Participants will have a baseline visit which will include repeat of the screening testing.

Participants will then present for their first study visit which will include: receiving vedolizumab infusions through an arm vein, repeats of the baseline testing. Participants will then have serial visits on a pre-specific schedule to receive ongoing vedolizumab doses every 2-4 weeks until week 20. Each visit will also include repeat of the baseline tests.

After week 6 and before week 7 patients will discontinue ART. After the final infusion of vedolizumab at week 20 patients will continue to be assessed with physical exam, medical history, and repeat of the baseline testing every 4 weeks up to 1 year.

ART will be re-started for participants if the level of HIV in the blood becomes too high, persists for too long, or if the CD4 count decreases by too much.

DETAILED DESCRIPTION:
HIV is a chronic active infection of lymphocytes and monocytoid cells resulting in a progressive and profound depletion of T cell subsets and ultimately in acquired immune deficiency syndrome (AIDS). HIV infects cells of the immune system throughout the body and may cause an active cytolytic infection in activated lymphocytes, become dormant as a latent infection in resting lymphocytes, or continue as a chronically active infection in macrophages. Continuous anti-retroviral drug treatment (ART) suppresses virus within the bloodstream and allows some degree of immune healing so as to permit near-normal health and life expectancy. However, interruption of ART is uniformly followed by rebound of viremia as a result of ongoing chronic active infection, and reactivation of latent infection. Successful ART requires daily medications indefinitely. There is an ongoing need for treatments which are more effective in the eradication of HIV. Counter to past expectations for cell-mediated immunity, broadly neutralizing monoclonal antibodies (nmAb) have been developed which show anti-HIV activity in vivo in reducing viremia (plasma virus load, PVL), and in slightly reducing recurrence of lasting PVL following analytical treatment interruption (ATI). Monoclonal antibody therapies against host cellular markers such as HIV co-receptors have been put forward as potential strategy in immunological treatment of HIV infection. If activated lymphocytes could be protected from cytolytic HIV infection in the presence of concurrent active HIV infection of other cells and tissues, then unperturbed potent acquired specific or innate immunity might confer lasting immunological remission of HIV infection.

This year, an unexpected finding of sustained remission of plasma viremia level (PVL) to below quantifiable assay limits in a rhesus macaque SIV infection model of AIDS was reported. The envelope of SIV (and HIV) appears to interact with α4β7 integrin, a lymphocyte homing receptor for trafficking to gut mucosal-associated lymphoid tissue (GALT) that was the target of mAb treatment in this study. This study showed that in animals treated with the mAb while discontinuing ART there was a diminished rebound and sustained remission of PVL, and less GALT associated viral load for a long-lasting period of at least 24 months. The mechanism of this unexpected post-treatment effect is unknown. In humans infected with HIV, such an effect sustained over time with continued remission of progressive immunodeficiency would meet definitional criteria of "functional cure" of HIV/AIDS. The results observed in the SIV model reveal a promising avenue for investigation in this area of research towards control of HIV infection in absence of ART. We propose to assess the safety and tolerability of anti-α4β7 integrin monoclonal antibody in healthy HIV-infected adults on ART, to assess the safety of ATI and whether anti-α4β7 integrin monoclonal antibody treatment can induce sustained virologic remission in the absence of ART.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 to 65 years) with HIV infection.
2. Nadir CD4 T cell count ≥ 200 and current CD4 T cell count > 500 cells/mcL
3. Adherent on ART 2 to 9 years with sustained pVL ≤ 50 copies/mL
4. Ability to comprehend and provided informed consent

Exclusion Criteria:

1. Past AIDS-defining or AIDS-related immune deficiency diseases
2. Past drug-resistant HIV or ART-refractory pVL response
3. Current hepatitis B or C virus infection, or untreated latent TB infection
4. Clinically significant concurrent health condition.
5. Pregnancy, lactation, or non-adherence with contraception if fertile.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Vedolizumab safety and tolerance | 6 months vedolizumab treatments, serial assessments over 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, with their timing of onset and resolution.

SECONDARY OUTCOMES:
PVL rebound and remission after ATI on vedolizumab treatment, and after discontinuation of vedolizumab. | serial phlebotomy measures over 12 months
  Quantitative PVL (Abbott HIV1 Viral Load Assay) measured serially during and after ATI.
PVL sustained rebound after ATI, and re-suppression on ART. | serial phlebotomy measures over 12 months
  Quantitative PVL (Abbott HIV1 Viral Load Assay) measured serially during and after ATI.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Cameron, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital -General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Study dataset, after study closure and publication, by request.

REFERENCES:
- [Derived] Barros PO, Burke Schinkel SC, Nayak AL, Haas B, Berthoud TK, McGuinty M, Cameron DW, Angel JB. Failure of gammadelta T Cell Recovery in the Gut With Effective Anti-HIV Therapy. J Immunol Res. 2025 Nov 27;2025:9883892. doi: 10.1155/jimr/9883892. eCollection 2025. PMID 41323021
- [Derived] McGuinty M, Angel JB, Cooper CL, Cowan J, MacPherson PA, Kumar A, Murthy S, Sy R, Dennehy M, Tremblay N, Byrareddy SN, Cameron DW. Vedolizumab treatment across antiretroviral treatment interruption in chronic HIV infection: the HAVARTI protocol for a pilot dose-ranging clinical trial to assess safety, tolerance, immunological and virological activity. BMJ Open. 2020 Oct 8;10(10):e041359. doi: 10.1136/bmjopen-2020-041359. PMID 33033101